CLINICAL TRIAL: NCT04704492
Title: An Open-label, Multiple-dose Study to Assess the Pharmacokinetics, Pharmacodynamics, Preliminary Clinical Activity and Safety of Human Mouse Chimeric Anti-CD22 Monoclonal Antibody (SM03) in Patients With Rheumatoid Arthritis
Brief Title: A Study of the Pharmacokinetics and Safety of SM03 in Patients With Rheumatoid Arthritis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: SinoMab BioScience Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SM03-RA(I/II)-1.0; CTR20131127 (Other: chinadrugtrials.org.cn)
Record Dates: First submitted 2021-01-06; First posted 2021-01-11 (Actual); Last update posted 2021-01-11 (Actual); Status verified 2021-01

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Biological: SM03 (Experimental): Biological: SM03 600 mg or 900 mg intravenous (IV) on week 0 , 2.
  Interventions: Drug: Biological: SM03

INTERVENTIONS:
Drug: Biological: SM03 — Biological: SM03 600 mg or 900 mg intravenous (IV) on week 0,2
  Other Names: SM03

SUMMARY:
This was an open phase I trial to evaluate the pharmacokinetic, pharmacodynamic, safety and clinical activity profiles of anti-CD22 monoclonal antibody SM03 in patients with active RA.

DETAILED DESCRIPTION:
This was an open phase I trial to evaluate the PK, PD, safety,tolerability, efficacy, and immunogenicity of SM03 in patients with RA. The total study duration was approximately 16 weeks for each participant, including a screening period of maximally 4 weeks, a multiple-dose period of 2 weeks (day 0 ~ day 14), and a post-treatment follow-up period of 10 weeks (day 15 ~ day 84).

ELIGIBILITY:
Inclusion Criteria:

* Rheumatoid arthritis (RA) for ≥ 6 months, diagnosed according to the revised 1987 American College of Rheumatology (ACR) criteria for the classification of rheumatoid arthritis.
* Moderate to severe active RA with swollen joint count (SJC) ≥ 6 (66 joint count), and tender joint count (TJC) ≥ 8 (68 joint count) at screening and baseline.
* At screening, either C-reactive protein (CRP) ≥ 0.6 mg/dL (6 mg/L), or Erythrocyte sedimentation rate (ESR) ≥ 28 mm/hour, or Morning stiffness of joint for ≥ 45 minutes.
* Receiving methotrexate (MTX) 7.5 - 25mg/week (oral) for at least 12 weeks, at a stable dose over the past 4 weeks.

Exclusion Criteria:

* Females who are pregnant, breastfeeding, or planning a pregnancy during the Treatment Period of and 12 months after the last infusion of study drug.
* Rheumatic autoimmune disease other than RA.
* Use of any biological DMARDs for RA within past 6 months.
* Active infection, or history of serious or chronic infection.
* Any significant cardiac disease, moderate to severe chronic obstructive pulmonary disease.
* Allergy or sensitivity to components of the drug vial or any of the materials used for infusion

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2012-08-14 (Actual); Primary Completion 2013-12-16 (Actual); Study Completion 2013-12-16 (Actual)

PRIMARY OUTCOMES:
Area Under the Concentration Time Cure(AUC0-t) | Week 0 to 12
  Pharmacokinetic endpoint: Area Under the Concentration Time Cure(AUC0-t)
Time to Maximum Plasma Concentration (Tmax) | Week 0,2
  Pharmacokinetic endpoint: Time to Maximum Plasma Concentration (Tmax)
Peak Plasma Concentration (Cmax) | Week 0, 2
  Pharmacokinetic endpoint: Peak Plasma Concentration (Cmax)
Systemic Clearance (CL) | Week 0 to 12
  Pharmacokinetic endpoint: Systemic Clearance (CL)
Terminal Half-life (T1/2) | Week 0 to 12
  Pharmacokinetic endpoint:Terminal Half-life (T1/2)

SECONDARY OUTCOMES:
Number of Participants Who Experienced at Least One Adverse Event | Week 0 to 12
  An adverse event is defined as any unfavorable and unintended sign including an abnormal laboratory finding, symptom or disease associated with the use of a medical treatment or procedure, regardless of whether it is considered related to the medical treatment or procedure.
Number of ACR20, ACR50, and ACR70 Responders at Week 12 | Week 2,4,8,12
  American College of Rheumatology (ACR) Responder Index is based on a set of evaluations: the Investigator Tender Joint Count/Number of Tender Joints (out of 68 Joints); Investigator Swollen Joint Count/Number of Swollen Joints (out of 66 Joints); Patient Global Assessment of Disease Activity (PGAD); Investigator Global Assessment of Disease Activity (IGAD); Patient Global Assessment of Pain (PGAP); Health Assessment Questionnaire Disability Index (HAQ-DI); and ESR. ACR response indicates percent change (ie, improvement) from baseline (20%, 50%, 70%) PGAD & IGAD
Change From Baseline in Disease Activity Score (DAS28-ESR) at Week 12 | Week 0,2,4,8,12
  The DAS28 is a composite score to measure disease activity in patients with rheumatoid arthritis, derived from the following variables:
  The number of swollen and tender joints assessed using the 28-joint count; Erythrocyte sedimentation rate (ESR); Patient's global assessment of disease activity measured on a 10 cm visual analog scale.
  The DAS28 score ranges from zero to ten. A DAS28 score above 5.1 means high disease activity whereas a DAS28 less than or equal to 3.2 indicates low disease activity. Remission is achieved by a DAS28 lower than 2.6.

OTHER OUTCOMES:
Number of Participants Positive for Anti-Drug Antibody (ADA) | Week 0,4,8,12
  Serum ADA positivity is determined over course of the trial duration
Change From Baseline in CD19+ B-cell Count During the Study Period | Week 0,4,8,12
  Pharmacodynamic endpoint: change from baseline in CD19+ B-cell count during the study period

CONTACTS AND LOCATIONS:
Overall Officials: Pei Hu, PhD,MD, Principal Investigator — Clinical Pharmacology Research Center & Translational Medicine Centre, Peking Union Medical College Hospital
Locations (1):
- Clinical Pharmacology Research Center & Translational Medicine Centre, Peking Union Medical College Hospital, Beijing, China